CLINICAL TRIAL: NCT00032760
Title: Meditation-Based Treatment for Binge Eating Disorder
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: R21AT000416-01 (NIH)
Record Dates: First submitted 2002-04-01; First posted 2002-04-02 (Estimated); Last update posted 2007-10-02 (Estimated); Status verified 2007-09

CONDITIONS: Binge Eating Disorder; Obesity
Keywords: binge eating disorder; human therapy evaluation; meditation; obesity; nutrition education; psychotherapy; racial /ethnic difference; adult human; alternative medicine; patient oriented research
MeSH Terms: conditions — Binge-Eating Disorder; Obesity | interventions — Meditation

INTERVENTIONS:
Behavioral: Meditation

SUMMARY:
The purpose of this study is to assess the relative effectiveness of a mindfulness meditation-based intervention for binge eating disorder in comparison to a psycho-educational intervention and a waiting-list control group.

DETAILED DESCRIPTION:
As many as 30% of individuals seeking treatment for obesity meet the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) criteria for binge eating disorder (BED). BED is marked by recurrent episodes of bingeing, accompanied by feelings of loss of control, and involves chronic disregulation of physiological, emotional and behavioral systems. Meditation-based interventions have been used successfully to treat disorders with similar addictive and disregulatory characteristics, but have not been applied to treating BED. Data from an uncontrolled pilot study suggests that such an intervention can have marked immediate impact on decreasing episodes of binge eating and other associated characteristics in obese women. Therefore, this study incorporates appropriate comparison conditions to further investigate the efficacy of a mindfulness meditation-based intervention as a treatment component for treating BED symptoms. Exploratory aspects include further development of a manual, establishment of effect size (in comparison to appropriate comparison groups), inclusion of a more diverse population, and of measures that address: 1) individual differences in treatment response, 2) possible mechanisms, 3) time course of response, and 3) impact on medical/health variables.

Women from two communities will be randomly assigned to 3 conditions: 1) an 8-week manualized meditation-based group intervention, 2) a psychoeducational comparison condition, or 3) a waiting-list control. Primary outcome variables will be changes in binge eating behaviors, and associated measures of depression, anxiety, self-esteem, and diet; secondary variables include medical variables sensitive to dietary change (i.e., weight; blood pressure; lipid profile; blood glucose levels), and process variables related to meditation practice, such as the Tellegen Absorption Scale, perceived value and use of the meditation practice, and experiences of increased control and awareness. Participants will be evaluated pre- and post-treatment, and at 1, 3, and 6 months followup. This data would then support the further investigation of a meditation-based intervention as part of a more comprehensive treatment program for BED.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of binge eating disorder;
* BMI at least 30;
* Fluent English speaker/reader;
* Able and willing to attend 9 weekly group sessions over two months, plus followup for 6 months, either in geographic area of Terre Haute, Indiana, or Durham, North Carolina.

Exclusion Criteria:

* Psychiatric or other condition that would preclude appropriate group participation;
* On a structured diet program;
* Unstable related medical syndrome (e.g., diabetes, hypertension);
* Medication that affects weight or appetite that is still being adjusted or that is likely to change during the course of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160
Dates: Start 2002-03; Study Completion 2004-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean L. Kristeller, PhD, Principal Investigator — Indiana State University; Ruth Quillian-Wolever, PhD, Principal Investigator — Duke University Department of Psychiatry/Center for Integrated Medicine
Locations (2):
- United States (2):
  - Indiana State University, Terre Haute, Indiana
  - Duke Center for Integrative Medicine, Durham, North Carolina

REFERENCES:
- [Background] Kristeller JL, Hallett CB. An Exploratory Study of a Meditation-based Intervention for Binge Eating Disorder. J Health Psychol. 1999 May;4(3):357-63. doi: 10.1177/135910539900400305. PMID 22021603